CLINICAL TRIAL: NCT06333015
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Study to Evaluate the Safety and Effectiveness of the enVista® Beyond (EY) EDF Intraocular Lens in Subjects Undergoing Cataract Extraction
Brief Title: Study to Evaluate the Safety and Effectiveness of the enVista® Beyond (EY) EDF Intraocular Lens in Subjects Undergoing Cataract Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 924
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Approximately 299 subjects will be randomized in the study. In the first phase 224 subjects will be randomized at a 1:1 ratio to either the test or control IOL, and in the second phase 75 subjects will be randomized at a 2:1 ratio to either the test or control IOL.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and designated postoperative evaluator(s) will be masked to the IOLs assigned. The Investigator implanting the IOL and designated site personnel will be unmasked to the treatment assignment for a subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- enVista Beyond EY IOL (Experimental): Subjects implanted with enVista Beyond Extended Depth of Focus (EDF) Intraocular Lens (IOL) Model EY
  Interventions: Device: enVista Beyond EY (EDF) IOL
- enVista MX60E monofocal IOL (Active Comparator): Subjects implanted with enVista MX60E monofocal IOL
  Interventions: Device: enVista MX60E monofocal IOL

INTERVENTIONS:
Device: enVista Beyond EY (EDF) IOL — enVista Beyond Extended Depth of Focus (EDF) Intraocular Lens (IOL) Model EY
  Arms: enVista Beyond EY IOL
Device: enVista MX60E monofocal IOL — enVista MX60E monofocal IOL
  Arms: enVista MX60E monofocal IOL

SUMMARY:
This research study is evaluating the safety and efficacy (performance) of the Bausch + Lomb enVista Beyond Hydrophobic Acrylic Extended Depth of Focus Intraocular Lens (IOL) in subjects who receive this IOL in both eyes.

DETAILED DESCRIPTION:
The study will evaluate the safety and effectiveness of the enVista Beyond (EY) EDF IOL in providing increased depth of focus, comparable distance and improved near and intermediate visual acuity compared to the parent enVista monofocal IOL. This is a prospective, multicenter, randomized, controlled, subject and visual acuity assessor masked, parallel-group study in subjects bilaterally implanted with either EY or enVista MX60E monofocal IOL following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 22 years of age or older on the date the Informed Consent Form (ICF) is signed.
2. Subjects must have the capability to understand and provide written informed consent on the Institutional Review Board (IRB) approved ICF and authorization as appropriate for local privacy regulations.
3. Subjects must have a BCDVA equal to or worse than 20/40 in each eye, with or without a glare source present (Brightness Acuity Tester), or have significant cataract-related visual symptoms, due to a clinically significant cataract (cortical, nuclear, subcapsular, or combination) that is considered amenable to treatment with standard phacoemulsification cataract extraction and capsular IOL implantation.
4. Subjects must have preoperative corneal astigmatism less than 1.0 D for each eye.
5. Subjects must have a BCDVA projected to be better than 20/30 after cataract removal and IOL implantation in each eye, as determined by the medical judgment of the Investigator or measured by potential acuity meter (PAM) testing, if necessary.
6. Subjects must have clear intraocular media other than the cataract in both eyes.
7. Contact lens wearers must demonstrate a stable refraction (within ±0.50 D in magnitude for both sphere and cylinder and within ±15° in axis) in both eyes, as determined by distance manifest refraction on two consecutive examination dates (both refractions performed at least 7 days apart) after discontinuation of contact lens wear (Rigid or Toric lenses discontinued for at least 2 weeks and soft contact lenses discontinued for at least 3 days prior to the first refraction used to establish stability and through the day of surgery).
8. Subjects must require an IOL power from +14.0 diopter (D) to +28.0 D for each eye.
9. Subjects must be willing and able to comply with all treatment and follow-up study visits and procedures, and to undergo second eye surgery within 7-30 days of the first eye surgery.

Exclusion Criteria:

1. Subjects who have used an investigational drug or device within 30 days prior to the planned first surgery date and/or will participate in another investigation during the period of study participation.
2. Subjects with presence of any corneal pathology (e.g., significant scarring, guttata, inflammation, edema, dystrophy, etc.), not including mild superficial punctate keratitis (SPK) (confirmed by corneal staining), in either eye.
3. Subjects with conditions that increase the risk of zonular rupture during cataract extraction procedure that may affect the postoperative centration or tilt of the lens.
4. Subjects who have uncontrolled glaucoma in either eye. Uncontrolled glaucoma is defined as intraocular pressure (IOP) greater than 21 mm Hg in spite of maximally tolerated medications (with more than 3 topical drugs for IOP control).
5. Subjects with previous retinal detachment or presence or history of clinically significant retinal pathology involving the macula in either eye.
6. Subjects with presence of proliferative or non-proliferative diabetic retinopathy in either eye.
7. Subjects who have a congenital ocular anomaly (e.g., aniridia, congenital cataract) in either eye.
8. Subjects using any systemic or topical drug known to interfere with visual performance, pupil dilation, or iris structure within 30 days of randomization (refer to the relevant attachment of the Study Reference Manual).
9. Subjects who have a history of chronic or recurrent inflammatory eye disease (e.g., iritis, scleritis, iridocyclitis, or rubeosis iridis) in either eye.
10. Subjects with presence or history of diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are expected to cause future visual acuity losses to a level of 20/30 or worse in either eye.
11. Subjects who have had previous intraocular or corneal surgery in either eye that might confound the outcome of the investigation or increase the risk to the subject.
12. Subjects with any active infectious conjunctivitis, keratitis, or uveitis in either eye.
13. Subjects who have irregular astigmatism or skewed radial axis for either eye.
14. Subjects who cannot achieve a minimum pharmacologic pupil dilation of at least 5.0 mm in both eyes.
15. Subjects who may be expected to require a combined or other secondary surgical procedure in either eye (note: corneal incisions intended specifically to reduce astigmatism are not allowed during the study).
16. Females of childbearing potential (those who are not surgically sterilized or at least 12 months postmenopausal) are excluded from the study if they are currently pregnant or plan to become pregnant during the study, lactating or have a condition associated with fluctuation hormones that could lead to refractive changes. Females of childbearing potential must be willing to practice effective contraception for the duration of their participation in the study.
17. Subjects with any other serious ocular pathology or underlying systemic medical disease (e.g., uncontrolled diabetes) or circumstance that, based on the Investigator's judgment, poses a concern for the subjects' safety, increases the operative risk or could confound the results of the study.
18. Subjects who have current or previous usage of systemic medications that may confound the outcome or increase the risk to the subject based on the Investigator's judgement. For example; subjects on an alpha-1-selective adrenoceptor blocking agent or an antagonist of alpha 1A adrenoceptor (e.g., tamsulosin hydrochloride (Flomax®), Terazosin, Rapaflo or Cardura) or other medications with similar side effects (floppy iris syndrome).
19. Subjects who are expected to require retinal laser treatment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean Monocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Monocular photopic DCIVA (logMAR) will be measured at 66 cm in the first implanted eye.
Median Monocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Monocular photopic DCIVA (logMAR) will be measured at 66 cm in the first implanted eye.
Negative lens induced distance-corrected Depth of focus (D) at 0.20 logMAR of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Negative lens induced distance-corrected Depth of focus (D) at 0.20 logMAR in the first implanted eye.
Mean monocular best-corrected distance visual acuity (BCDVA) (logMAR) of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Monocular Photopic Best-Corrected Distance Visual Acuity (BCDVA) (logMAR) will be measured at 4 meters in the first implanted eye.
Rates with postoperative monocular BCDVA of 20/40 (0.30 logMAR) or better of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Rates with postoperative monocular BCDVA of 20/40 (0.30 logMAR) or better in the first implanted eye. Monocular Photopic Best-Corrected Distance Visual Acuity (BCDVA) (logMAR) will be measured at 4 meters.

SECONDARY OUTCOMES:
Mean monocular photopic distance-corrected near visual acuity (DCNVA) of first implanted eyes at Post-Operative Visit 4. | Day 120 to Day 180 after second eye implantation
  Monocular photopic DCNVA (logMAR) will be measured at 40 cm in the first implanted eye.

CONTACTS AND LOCATIONS:
Overall Officials: Rosangela Sonner, Study Director — Bausch & Lomb Incorporated
Locations (16):
- United States (16):
  - Site 119, Dothan, Alabama
  - Site 108, Northridge, California
  - Site 116, Alexandria, Minnesota
  - Site 107, Bloomington, Minnesota
  - Site 101, Omaha, Nebraska
  - Site 109, Las Vegas, Nevada
  - Site 113, Garden City, New York
  - Site 118, West Fargo, North Dakota
  - Site 102, Brecksville, Ohio
  - Site 105, North Charleston, South Carolina
  - Site 106, Sioux Falls, South Dakota
  - Site 103, Dallas, Texas
  - Site 117, San Antonio, Texas
  - Site 112, San Antonio, Texas
  - Site 115, Sugar Land, Texas
  - Site 111, Mount Pleasant, Wisconsin

IPD SHARING:
Plan to Share IPD: No